CLINICAL TRIAL: NCT05655936
Title: Eliminating Severe Maternal Morbidity With Heart Health Doulas Trial
Acronym: HHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Janet Catov, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY22060056; 1R01MD017083-01A1 (NIH)
Record Dates: First submitted 2022-12-08; First posted 2022-12-19 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-05

CONDITIONS: Preeclampsia; Hypertensive Disorder of Pregnancy; Toxemia; Pregnancy Complications; Hypertension, Pregnancy-Induced; Hypertension; Obesity; Overweight; Nutrition Disorders; Vascular Diseases; Cardiovascular Diseases; Pre-Eclampsia; Eclampsia; Gestational Hypertension
Keywords: Postpartum Doula, Doula Intervention
MeSH Terms: conditions — Pre-Eclampsia; Toxemia; Pregnancy Complications; Hypertension, Pregnancy-Induced; Hypertension; Obesity; Overweight; Nutrition Disorders; Vascular Diseases; Cardiovascular Diseases; Eclampsia

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a prospective single site, single-blinded, parallel randomized control trial in which women diagnosed with HDP will be randomized into either the control or intervention group. The investigators will randomize 454 women into usual care, or an 8-12-week heart health intervention program provided by a postpartum Doula. Randomization will be stratified by race to achieve over enrollment of Black and African American participants.
Who Masked: Participant
Masking Description: Participants and Investigators will be blinded until randomization assignment is executed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Group (Active Comparator): The usual care group will receive remote blood pressure monitoring for approximately 6 weeks via the clinical home blood pressure monitoring program at Magee Women's Hospital of UPMC and be discharged after delivery as usual. This monitoring is standardly offered to women post-delivery with hypertensive disorders of pregnancy. Participants will text in their blood pressures to the medical record systems and be monitored by clinical staff.
  Interventions: Behavioral: Usual Care
- Postpartum Doula Intervention Group (Experimental): The intervention group will receive study devices (blood pressure cuff, scales, etc.) and instructions on 10-12 months of remote blood pressure, and weight monitoring. An electronic referral will be sent to the Healthy Start program to initiate postpartum Doula support for 8-12 weeks, and a Doula moderated social support group for 6 months. The postpartum Doula will deliver a heart health focused intervention aimed at reducing blood pressure by approximately 12 weeks postpartum.
  Interventions: Behavioral: Heart Health Doula Intervention Program; Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Heart Health Doula Intervention Program — The intervention group will be given a smart blood pressure cuff and a smart scale to monitor weight. The intervention group will receive support provided a postpartum doula until 8-12 weeks postpartum. The doula will provide individualized support during this time, and after 8-12 weeks, women will transition to a doula-moderated support group for the remainder of the study. The intervention group will continue to receive blood pressure and weight monitoring for the remainder of the study.
  Arms: Postpartum Doula Intervention Group
Behavioral: Usual Care — Usual care includes enrollment into a clinical 6-week home-based blood pressure monitoring program with text messaging support which includes receiving a home blood pressure cuff. Women in the intervention group will be offered the same support as the usual care group, and in addition will receive the intervention and supplies.

SUMMARY:
This is a single site, single-blinded parallel randomized control trial that investigates a multi-level intervention to improve postpartum blood pressure in women with hypertensive disorder pregnancy. The investigators will recruit women diagnosed with a hypertensive disorder of pregnancy, identified between 3rd trimester and 2 weeks post-delivery. The investigators will randomize participants to receive usual care home blood pressure monitoring for 6 weeks versus an intervention of usual care + blood pressure and weight monitoring + a doula trained in heart health. This trial will be conducted in partnership with a local community-based organization, Healthy Start Inc.

DETAILED DESCRIPTION:
The purpose of this study is to improve blood pressure in women who have a hypertensive disorder of pregnancy. A hypertensive disorder of pregnancy is one in which a woman's blood pressure is elevated during pregnancy. For the purpose of this project, a hypertensive disorder of pregnancy includes gestational hypertension, preeclampsia and eclampsia. By improving blood pressure in pregnant women, the investigators aim to lower the number of women with chronic hypertension, cardiovascular disease, and mortality. The study will enroll 454 women who are 18 years or older, are about to or have recently given birth, and have been diagnosed with a hypertensive disorder of pregnancy. Women will be randomly chosen to take part in usual care or an intervention group.

This study is designed to evaluate support for new moms by providing a postpartum doula in partnership with Healthy Start Inc. Healthy Start is a local community-based organization that supports women, children, fathers, families and communities through community-based programming, advocacy, research, and training. The support provided to new moms will include weekly doula sessions (in-person or virtual), education and support, and blood pressure and weight monitoring. Women will be enrolled during their third trimester up until they are a few weeks postpartum and will complete the study around 12 months postpartum. If assigned to the intervention group, women will attend weekly check-ins with their doula for 8-12 weeks and receive continuous blood pressure and weight monitoring throughout the duration of the study. Both groups will be enrolled into a 6-week home-based blood pressure monitoring program with text messaging support (enrollment in the 6-week program is the standard of care at Magee Women's Hospital following a hypertensive disorder of pregnancy). Both the usual care and intervention groups will attend a follow-up visit at 12 months postpartum.

ELIGIBILITY:
Inclusion

* Women must be pregnant or postpartum and assessed during pregnancy and/or delivery with a diagnosis of a hypertensive disorder of pregnancy (pre-eclampsia, eclampsia or gestational hypertension).
* Women must reside in Allegheny, Westmoreland, Beaver, Butler, or Washington County. Participant may also reside within 100 miles of Allegheny County.
* The participant must deliver (or plan to deliver) at Magee-Womens Hospital

Exclusion

* No pre-pregnancy chronic conditions that affect blood pressure such as hypertension or on antihypertensive medications within 3 months before conception.
* No diabetes (type 1 or type 2)
* No chronic and severe renal or liver disease or systemic lupus erythematous
* No women under the age of 18

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Assess MAP at 12 months postpartum | Baseline to approximately 12 months postpartum
  To test the effectiveness of the postpartum Doula intervention the investigators will evaluate blood pressure and mean arterial pressure (MAP) at 12 months postpartum.

SECONDARY OUTCOMES:
Change from baseline in racial disparities and blood pressure & MAP at 12 months | Baseline to approximately 12 months postpartum
  To determine if an enhanced care strategy reduces racial disparities in blood pressure, the investigators will evaluate blood pressure and mean arterial pressure (MAP) recovery by 12 months postpartum by race and by intervention group. Systolic and diastolic blood pressures will be assessed separately. There is evidence that blood pressure should normalize at 6-12 months postpartum and by assessing black vs white differences, the investigators will determine if the intervention can reduce known disparities in blood pressure and MAP.
Assess Racial Disparities in Healthcare Delivery | Up to 12 months postpartum
  Access to optimal clinical care is essential for all women to successfully recover from a hypertensive disorder of pregnancy (HDP) within one year postpartum. The investigators will assess racial differences in healthcare service delivery that contribute to inequities in HDP-related care by reviewing the charts of women who enroll in the study and comparing whether care was received, and the type of care aligned with the guidelines/standards by indicating whether the care met, did not meet, or exceeded the standards at critical time points.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Catov, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Magee Women's Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data (including data dictionaries) will be shared at the direction of the primary investigator. Data will include blood pressure, weight, demographics, physical activity, and pregnancy related information. Additional documents (such as the study protocol) will be made available. The dataset for our project will be prepared according to requirements for and stored on the Clinicaltrials.gov data repository. Per the NIH guidelines, the dataset will be submitted to the program officer within a year after the outcomes are published and no later than 3 years after the end of clinical activities.
Supporting Information: Study Protocol
Time Frame: Within a year after outcomes are published and no later than 3 years after the end of clinical activities.
Access Criteria: NHLBI data repository request process
URL: https://biolincc.nhlbi.nih.gov/home/